CLINICAL TRIAL: NCT03305484
Title: Contact Lens Assessment in Youth - Soft Contacts Observation of Risk and Education (CLAY-SCORE)
Brief Title: Soft Contacts Observation of Risk and Education (SCORE)
Acronym: SCORE
Status: Completed | Type: Observational
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: University of Houston (Other); New England College of Optometry (Other); Ohio State University (Other); University of Waterloo (Other); Pacific University (Other); Nova Southeastern University (Other); Alcon Research (Industry)
Responsible Party: Principal Investigator, Dawn Lam, MSc, OD, Associate Professor, Southern California College of Optometry at Marshall B. Ketchum University
Other Study IDs: SCCO-16-15; IIT#23485303 (Other Grant/Funding Number: Alcon)
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Contact Lens Complication; Contact Lens Acute Red Eye; Contact Lens Related Corneal Infiltrate (Disorder); Contact Lens-Induced Corneal Fluorescein Staining
Keywords: contact lenses; red eye; corneal infiltrate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic Contact Lens Wearers: Contact lens wearers who present to the eye care practitioner's office with a symptomatic red eye
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, observation only
  Other Names: No intervention, observation only

SUMMARY:
Specific Aims

1. Develop risk assessment scores for SCL wearers
2. Test the scoring algorithm in SCL wearers who present with adverse events
3. Explore targeted patient education to reduce risk behaviors associated with SCL wear.

DETAILED DESCRIPTION:
This will be a multi-center, case-control prospective study. Subjects will be enrolled at five geographically diverse locations across North America. The intent is to enroll cases with new (untreated) red eyes and controls that are representative of the contact lens wearing population and test the new scoring algorithm on this population.

A total of 232 participants are expected to complete the study (116 case-control sets). Enrollment will be competitive. After consent, subjects will complete the Contact Lens Risk Survey (CLRS) online at www.claystudy.org. Data related to symptoms, medical history and anterior segment evaluation will be collected. Subjects will be treated as usual and customary by the investigator. No intervention of treatment in this study. Subjects will be asked to repeat the CLRS at one and six months post initial visit.

Initial factor analysis from the previous CLRS data were used to develop and test the CLRS algorithm. Five sub-scales were identified in the areas of contact lens care, contact lens dependence, hygiene, living arrangements and wellness. Assuming a 10% missing data rate, a total of 58 SCL wearers with "serious and significant" red eye events will allow for detection of 0.4 or larger effect size.

There are multiple steps to "compliant wear" of contact lenses and while many patients do many of the correct wear behaviors, it's not realistic for practitioners to re-educate all wearers on all of the steps necessary to successfully wear SCLs. The CLRS allows patients to quickly report their specific wear behaviors and then receive only the targeted information on which behaviors they are doing that puts them at higher risk. A previous CLAY study demonstrated good repeatability of the CLRS survey one week after initial fielding.

ELIGIBILITY:
Inclusion Criteria:

* CASES

  * Current SCL wear (as defined by having worn lenses in previous week) without restriction on lens material, design, indication, wearing schedule or lens power
  * 18 - 39 years of age
  * New (untreated) symptomatic red eye CONTROLS
  * Current SCL wear (as defined by having worn lenses in previous week) without restriction on lens material, design, indication, wearing schedule or lens power
  * 18 - 39 years of age and gender and age-matched (± 3 years) to Case
  * Have not had an eye care examination within the past three months

Exclusion Criteria:

* CASES

  * Faculty, staff or student at an optometry college or school
  * Family or household member of an eye care provider, ophthalmic technician, ophthalmology or optometry residents or optometry students
  * Pregnancy (by self-report)
  * Currently enrolled in another eye/vision clinical trial
  * Previous participant in a CLAY study
  * Wearing SCL in conjunction with gas permeable (GP) lenses (i.e., piggyback design, hybrid lens.) CONTROLS
  * Same exclusion criteria as cases

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: A total of 232 participants are expected to complete the study (116 case-control sets). Enrollment will be competitive; with each of five geographic locations in the United States and Canada enrolling approximately 24, but no more than 29 case-control sets until the total sample size of is achieved.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Validation of the Contact Lens Risk Survey (CLRS) | twelve months
  This study will further validate the CORS and facilitate its translation into clinical practice. A scoring algorithm will be developed.
Targeted Patient Education | twelve months
  Scripted patient education will be generated based on the results of the Contact Lens Risk Survey (CLRS) to determine if changes in behavior at the one and six month time point

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Lam, Principal Investigator — Marshall B. Ketchum University
Locations (5):
- United States (4):
  - Marshall B. Ketchum University, Fullerton, California
  - Nova Southeastern University College of Optometry, Fort Lauderdale, Florida
  - The Ohio State, College of Optometry, Columbus, Ohio
  - University of Houston, College of Optometry, Houston, Texas
- University of Waterloo, Optometry and Vision Science, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD